CLINICAL TRIAL: NCT02487251
Title: Effectiveness of Differing Levels of Support for Family Mealtimes on Obesity Prevention Among Head Start Preschoolers
Brief Title: Effectiveness of Differing Levels of Support for Family Mealtimes on Obesity Prevention Among Head Start Preschools
Acronym: SimplyDinner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Holly Brophy-Herb, Professor, Michigan State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-68001-23239
Record Dates: First submitted 2015-06-13; First posted 2015-07-01 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Obesity
Keywords: Obesity; Family Mealtimes; Prevention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental: Phase 1 Usual Exposure (Experimental): Participants receive no additional information about healthy eating, family mealtimes, nutrition education or meal planning beyond any usual coverage of these areas.
  Interventions: Behavioral: Usual Exposure
- Experimental: Phase 1 Mealtime support activities (Experimental): Participants will engage in mealtime support activities such as healthy eating classes, cooking demonstrations, provision of cookware, receipt of mealtime ingredients, receipt of prepared meals, make and eat meals).
  Interventions: Behavioral: Mealtime Supports
- Experimental: Phase 2- Usual Exposure (Experimental): Participants receive no additional information about healthy eating, family mealtimes, nutrition education or meal planning beyond any usual coverage of these areas.
  Interventions: Behavioral: Usual Exposure
- Experimental: Phase 2- Meal Delivery and Receipt of Cookware (Experimental): Participants will receive two prepared meals weekly for 12 weeks and will receive a comprehensive set of cookware
  Interventions: Behavioral: Mealtime Supports

INTERVENTIONS:
Behavioral: Mealtime Supports — Participants will receive or engage in a variety of supports for family mealtimes in Phase 1 (e.g., receipt of prepared meals, receipt of cookware, informational supports, classes). In Phase 2 of the study participants received two prepared meals per week for 12 weeks and received a comprehensive set of cookware at the beginning of the intervention period.
  Arms: Experimental: Phase 1 Mealtime support activities; Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Behavioral: Usual Exposure — Participants receive no supplemental information on family mealtimes beyond what is already currently received
  Arms: Experimental: Phase 1 Usual Exposure; Experimental: Phase 2- Usual Exposure

SUMMARY:
Socioeconomic disparities in early childhood place low-income children at 1.5 to 2 times higher risk for obesity compared to middle- to upper-income children. Obesity interventions have turned toward the promotion of family mealtimes. This study will test the effects of 6 intervention components reflecting differing levels of supports to ultimately reduce childhood obesity prevalence and increase the frequency of healthy family mealtimes and improve dietary quality. The investigators will test 6 intervention components in Phase 1 (Screening Phase), resulting in the implementation and evaluation via a randomized controlled trial of a "final" intervention model in Phase 2 (Confirming Phase). The investigators hypothesize that providing low-income families with effective supports to enhance family capability to plan and implement family mealtimes will lead to improvements in children's adiposity indices, dietary quality and frequency of family meals.

DETAILED DESCRIPTION:
This study is comprised of two phases. In the first phase of the study, we will test associations between participation in combinations of 6 intervention components reflecting differing levels of practical resources to increase the frequency of healthy family mealtimes, improve children's dietary quality and ultimately reduce childhood obesity prevalence. Phase 1 utilizes the Multiphase Optimization Strategy (MOST) design to test combinations of the 6 intervention components which include: (1) Meal Delivery: the home delivery of pre-made healthy family meals including recipes weekly (2) Ingredient Delivery: the home delivery of ingredients and recipes to make healthy family meals weekly; (3) Community Kitchen: community kitchen sessions in which families prepare healthy meals with recipes to take home weekly; (4) Didactics: nutrition education classes using the Preschool Obesity Prevention Series (POPS) curriculum (5) Cooking Lessons: cooking lessons/demonstrations with recipes weekly; and (6) Cookware/Flatware: delivery of flatware/ cookware to utilize for family meals delivered at the beginning of the intervention. The goal of Phase 1 is to identify the intervention components most robustly related to decreased BMI z-score, increased dietary quality and frequency of family meals. Phase 1 will enroll approximately 500 parents of preschoolers. The goal of Phase 2 is to test the selected intervention components (identified in Phase 1) in a randomized controlled trial with approximately 250 participants. Participants in both phases will be enrolled through Head Start programs and/or university research recruitment platforms, social media, and posted flyers. The intervention period in Phase 1 will be 8 weeks, and the intervention period in Phase 2 will be expanded to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Preschool aged child

Exclusion Criteria:

* Significant feeding/eating disorders that would preclude participation in the interventions
* Child is a foster child
* Parent is non-English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly E. Brophy-Herb, Ph.D., Principal Investigator — Michigan State University
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Jackson Community Action Agency Head Start, Jackson, Michigan
  - Capital Are Community Services Head Start, Lansing, Michigan

REFERENCES:
- [Derived] Kerver JM, Brophy-Herb HE, Sturza J, Horodynski MA, Contreras DA, Stein M, Garner E, Hebert S, Williams JM, Kaciroti N, Martoccio T, Van Egeren LA, Choi H, Martin CK, Mitchell K, Dalimonte-Merckling D, Jeanpierre LA, Robinson CA, Lumeng JC. Supporting family meal frequency: Screening Phase results from the Simply Dinner Study. Appetite. 2022 Jul 1;174:106009. doi: 10.1016/j.appet.2022.106009. Epub 2022 Mar 22. PMID 35337884
- [Derived] Brophy-Herb HE, Horodynski M, Contreras D, Kerver J, Kaciroti N, Stein M, Lee HJ, Motz B, Hebert S, Prine E, Gardiner C, Van Egeren LA, Lumeng JC. Effectiveness of differing levels of support for family meals on obesity prevention among head start preschoolers: the simply dinner study. BMC Public Health. 2017 Feb 10;17(1):184. doi: 10.1186/s12889-017-4074-5. PMID 28187722

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrollment across the study reflect the number of parent-child dyads enrolled. Data were collected from both parent and child. Baseline characteristics of child and parent age, ethnicity, and BMIz, are reported.
Period: Overall Study
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Started (Sample sizes reflect parent-child dyads enrolled in each study arm. The sample size for dyads equals that number of parents and that number of children. Among those who started per arm: 434 parents/434 children (Phase 1 Usual Exposure); 65 parents/65 children (Phase 2 Mealtime Support Activities); 152 parents/152 children (Phase 2 Usual Exposure); 159 parents/159 children (Phase 2 Meal Delivery and Receipt of Cookware).) | 434 | 65 | 152 | 159
Completed (Sample sizes reflect parent-child dyads enrolled in each study arm. The sample size for dyads equals that number of parents and that number of children. Among those who completed per arm: 366 parents/366 children (Phase 1 Usual Exposure); 55 parents/55 children (Phase 2 Mealtime Support Activities); 125 parents/125 children (Phase 2 Usual Exposure); 134 parents/134 children (Phase 2 Meal Delivery and Receipt of Cookware).) | 366 | 55 | 125 | 134
Not Completed | 68 | 10 | 27 | 25

BASELINE CHARACTERISTICS:
Population: Parents and preschool aged children; the numbers reported reflect dyads enrolled in each study arm. Phase 1 Usual Care = 434 parents/434 children; Phase 1 Mealtime Support Activities = 65 parents/65 children; Phase 2 Usual Care = 152 parents/152 children; Phase 2 Meal Delivery and Receipt of Cookware = 159 parents/159 children. Child and parent sex, age, ethnicity, child BMIz and parent BMI are reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware | Total
Number analyzed (Participants) | 434 | 65 | 152 | 159 | 810
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of child at study enrollment Population: Note that the number analyzed may differ from the total number enrolled due to missing data.
  years
    number analyzed (Participants) | 431 | 63 | 146 | 152 | 792
    (all) | 4.07 (.63) | 4.02 (.61) | 4.32 (.70) | 4.38 (.76) | 4.17 (.68)
Age, Continuous [Mean (Standard Deviation); unit: years] — This is the age of the parent at study enrollment.
  years | 30.0 (6.9) | 28.7 (5.6) | 33.9 (5.8) | 34.0 (5.8) | 31.65 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants] — This is the sex of the child.
  Participants
    Female | 220 | 25 | 75 | 89 | 409
    Male | 214 | 40 | 77 | 70 | 401
Sex: Female, Male [Count of Participants; unit: Participants] — This is the sex of the parent.
  Participants
    Female | 416 | 59 | 139 | 147 | 761
    Male | 18 | 6 | 13 | 12 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This is the ethnicity of the child as reported by the parent. Population: Note that the number analyzed may differ from the total number enrolled due to missing data.
  Participants
    Hispanic or Latino | 49 | 8 | 17 | 19 | 93
    Not Hispanic or Latino | 385 | 57 | 135 | 138 | 715
    Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This is the ethnicity of the parent.
  Participants
    Hispanic or Latino | 36 | 5 | 15 | 14 | 70
    Not Hispanic or Latino | 398 | 60 | 136 | 144 | 738
    Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Child BMIz [Mean (Standard Deviation); unit: zscore] — Child BMIZ at study enrollment; The z-score is based on United States Centers for Disease Control growth references for children. A z-score of 0 reflects the 50th percentile based on the US CDC children's reference growth charts. A z-score < -1.645 indicates that the child is underweight. A healthy BMIz score is between -1.645 and 1.036. BMIz >1.036 = criteria for overweight; BMIz >1.645 = criteria for obese Population: Please note that the sample sizes for data differ depending on the measure. For example, some BMIz data are missing in Phase 1 if the child was not home during the data collection visit to measured and measurements could not be obtained at other settings (e.g., at school). BMIz data are also missing extensively in Phase 2 due to the COVID-19 pandemic because in person data collection was not possible.
  zscore
    number analyzed (Participants) | 403 | 63 | 114 | 112 | 692
    (all) | .64 (1.07) | .72 (1.10) | .34 (1.03) | .40 (1.04) | .56 (1.07)
Parent BMI [Mean (Standard Deviation); unit: mean] — This is the body mass index of the parent at study enrollment. CDC guidelines note the following classifications: BMI <18.5 = underweight range; BMI 18.5 to <25 = healthy weight range; BMI 25.0 to < 30 = overweight range; BMI 30.0 or greater =obesity range.
  Please note that the sample sizes for data differ depending on the measure. For example, BMIz data are missing extensively in Phase 2 due to the COVID-19 pandemic because in person data collection was not possible.
  mean | 31.51 (13.96) | 30.44 (8.50) | 29.75 (13.30) | 29.85 (8.63) | 30.39 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Change in BMIz
Description: Research staff measured children without shoes or heavy clothing. Measures were taken twice and averaged. BMI was calculated and child BMIz derived. Child obesity was defined as BMI > 95th percentile and overweight/obesity defined as a BMI > 85th percentile for age and sex. Note that due to the COVID-19 pandemic, data on BMIz were not collected beginning in March 2020.
  The z-score is based on United States Centers for Disease Control growth references for children. A z-score of 0 reflects the 50th percentile based on the US CDC children's reference growth charts. A z-score < -1.645 indicates that the child is underweight. A healthy BMIz score is between -1.645 and 1.036. BMIz >1.036 = criteria for overweight; BMIz >1.645 = criteria for obese
Time Frame: Prior to the implementation of the intervention (Baseline) and immediately post the 12 week intervention period (Post).
Population: Preschool aged children
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Number analyzed (Participants) | 403 | 63 | 114 | 112
z-score | .0060 (.39) | .00027 (.37) | .04 (.44) | -.02 (.38)
Statistical Analysis 1: Comparison: Experimental: Phase 1 Usual Exposure vs Experimental: Phase 1 Mealtime Support Activities vs Experimental: Phase 2- Usual Exposure vs Experimental: Phase 2- Meal Delivery and Receipt of Cookware; We tested change in BMIz for each of the four study arms/groups; Test type: Equivalence — Phase 1 sought to determine effect sizes. For Phase 2, sample size was set at 125 per arm which, with 20% attrition, would enable detection of small to medium effect sizes of d = 0.40SD for continuous outcomes and 38% relative risk reduction for binary outcomes with a power of 80% and α = .05; p = .34, Mixed Models Analysis — p < .05 reflects the threshold for statistical significance. The calculated p value for change in BMIz is p = .34; Mean Difference (Final Values) = -0.15 — The reported estimation parameter is the effect size (cohen's d) for the change in BMIz (particularly in the Phase 2 sample)

2. Secondary Outcome: Change in Dietary Quality-Observed Fruit
Description: Report of the child's usual eating habits (fruit) using the Pennington Remote Food Photography method. When using the RFPM and SmartIntake app, parents place a reference card next to the child's food and capture images of the food selection and plate waste. The parent identifies foods that are not easily identified by wrappers or containers by typing a food description into a text box. These data and food images are automatically sent by the app to the server-based Food Photography Application©, which is used to manage the data collection process and analyze the food images to estimate energy and nutrient intake. First, the foods in the images were linked to a match from the United States Department of Agriculture's Food and Nutrient Database for Dietary Studies (FNDDS; USDA, 2018). Second, a standard portion image, which contains an image of the same or a similar food that was carefully weighed to represent various portion sizes, was identified from an archived food image database.
Time Frame: Prior to the implementation of the intervention (Baseline) and immediately post the 12 week intervention period (Post).
Population: Parents of preschool aged children; note that observed dietary quality data was only collected in Phase 2.
Measure: Mean (Standard Deviation); unit: cup equivalent
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Number analyzed (Participants) | 0 | 0 | 104 | 107
cup equivalent |  |  | -.03 (.26) | -.04 (.27)
Statistical Analysis 1: Comparison: Experimental: Phase 2- Usual Exposure vs Experimental: Phase 2- Meal Delivery and Receipt of Cookware; We tested change in observed fruit intake for each of the two study arms/groups in Phase 2 and compared change between the usual care and intervention groups; Test type: Equivalence — Sample size was set at 125 per arm which, with 20% attrition, would enable detection of small to medium effect sizes of d = 0.40SD for continuous outcomes and 38% relative risk reduction for binary outcomes with a power of 80% and α = .05. Phase 2 analyses included mixed modeling. Negative mean change values reflect a decrease in intake; positive values reflect an increase; p = .62, Mixed Models Analysis — p < .05 reflects the threshold for statistical significance. The calculated p value for change in observed fruit intake is p = .62; Mean Difference (Final Values) = -.07 — The reported estimation parameter is a standardized mean difference between the groups, specifically cohen's d

3. Secondary Outcome: Change in Dietary Quality- Observed Vegetables
Description: Report of the child's usual eating habits (fruit) using the Pennington Remote Food Photography Method
Time Frame: Prior to the implementation of the intervention (Baseline) and immediately post the 12 week intervention period (Post).
Population: Parents of preschool aged children. Note that observed dietary quality was not included in Phase 1.
Measure: Mean (Standard Deviation); unit: cup equivalent
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Number analyzed (Participants) | 0 | 0 | 104 | 107
cup equivalent |  |  | -.01 (.13) | .05 (.15)
Statistical Analysis 1: Comparison: Experimental: Phase 2- Usual Exposure vs Experimental: Phase 2- Meal Delivery and Receipt of Cookware; We tested pre to post change in observed vegetable intake for each of the two study arms/groups in Phase 2 and compared change between the usual care and intervention groups. Positive Observed dietary quality data was not collected in Phase 1; Test type: Equivalence — Sample size was set at 125 per arm which, with 20% attrition, would enable detection of small to medium effect sizes of d = 0.40SD for continuous outcomes and 38% relative risk reduction for binary outcomes with a power of 80% and α = .05; p = .009, Mixed Models Analysis — p < .05 reflects the threshold for statistical significance. The calculated p value for change in observed vegetable intake is p = .009; Mean Difference (Final Values) = .40

4. Secondary Outcome: Change in Dietary Quality-Parent Reported Fruit Intake
Description: Report of the child's usual eating habits using the Block Kids 2004 Food Frequency. Parents self-reported their children's dietary intake using the Block Dietary Data Systems Kids Food Screener-Last Week (BKFS, Version 2), a 41-item survey assessing nutrients and food groups in children aged 2-17 years (Hunsberger et al., 2015). Nutrients and food groups are reported from multiple items summed from each survey construct. The current study operationalized dietary quality in cup equivalent as reflecting the following food groupings as indicators of higher quality dietary patterns (Haya et al., 2013): fruit/fruit juice
Time Frame: Prior to the implementation of the intervention (Baseline) and immediately post the 12 week intervention period (Post).
Population: Parents of preschool aged children
Measure: Mean (Standard Deviation); unit: cup equivalent
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Number analyzed (Participants) | 355 | 52 | 125 | 125
cup equivalent | -.04 (.86) | .09 (1.01) | -.21 (.71) | -.10 (.73)
Statistical Analysis 1: Comparison: Experimental: Phase 1 Usual Exposure vs Experimental: Phase 1 Mealtime Support Activities vs Experimental: Phase 2- Usual Exposure vs Experimental: Phase 2- Meal Delivery and Receipt of Cookware; We tested pre to post change in parent reported child fruit intake for each of the four study arms/groups; Test type: Equivalence — Phase 1 sought to determine effect sizes. For Phase 2, sample size was set at 125 per arm which, with 20% attrition, enabled detection of small-medium effect sizes, d = 0.40SD for continuous outcomes and 38% relative risk reduction for binary outcomes, power of 80%, α = .05. Phase 1 analyses included paired t-tests & examination of pre-post effect size change. Phase 2 analyses included mixed modeling. Negative mean change values reflect a decrease in intake; positive values reflect an increase; p = .21, Mixed Models Analysis — p < .05 reflects the threshold for statistical significance. The calculated p value for change in parent reported fruit is p = .21; Mean Difference (Final Values) = .15 — The reported estimation parameter is a standardized mean difference between the groups, specifically cohen's d

5. Secondary Outcome: Change in Dietary Quality-Parent Reported Vegetables
Description: Parents self-reported their children's dietary intake using the Block Dietary Data Systems Kids Food Screener-Last Week (BKFS, Version 2), a 41-item survey assessing nutrients and food groups in children aged 2-17 years (Hunsberger et al., 2015). Nutrients and food groups are reported from multiple items summed from each survey construct. The current study operationalized dietary quality in cup equivalent as reflecting the following food groupings as indicators of higher quality dietary patterns (Haya et al., 2013): vegetables excluding potatoes and legumes.
Time Frame: Prior to the implementation of the intervention (Baseline) and immediately post the 12 week intervention period (Post).
Population: Parents of preschool aged children
Measure: Mean (Standard Deviation); unit: cup equivalent
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Number analyzed (Participants) | 355 | 52 | 125 | 125
cup equivalent | -.02 (.37) | .04 (.35) | -.06 (.30) | -.04 (.29)
Statistical Analysis 1: Comparison: Experimental: Phase 1 Usual Exposure vs Experimental: Phase 1 Mealtime Support Activities vs Experimental: Phase 2- Usual Exposure vs Experimental: Phase 2- Meal Delivery and Receipt of Cookware; We tested change in vegetable intake for each of the four study arms/groups; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = .55, Mixed Models Analysis — p < .05 reflects the threshold for statistical significance. The calculated p value for change in parent reported vegetables is p = .55; Mean Difference (Final Values) = .07 — The reported estimation parameter is a standardized mean difference between the groups, specifically cohen's d

6. Secondary Outcome: Change in Frequency of Healthy Family Mealtimes
Description: Using a 1-item question, parents reported how many nights in the week the parent and focus child are dinner together in the same place at home (e.g., in the kitchen) at the same time for most of the meal.
Time Frame: Prior to the implementation of the intervention (Baseline) and immediately post the 12 week intervention period (Post).
Population: Parents of preschool aged children
Measure: Mean (Standard Deviation); unit: mealtimes
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
Number analyzed (Participants) | 348 | 53 | 125 | 135
mealtimes | .08 (2.16) | .40 (2.29) | -.11 (1.95) | -.15 (1.56)
Statistical Analysis 1: Comparison: Experimental: Phase 1 Usual Exposure vs Experimental: Phase 1 Mealtime Support Activities vs Experimental: Phase 2- Usual Exposure vs Experimental: Phase 2- Meal Delivery and Receipt of Cookware; We tested change in frequency of family mealtimes for each of the four study arms/groups; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .84, Mixed Models Analysis — p < .05 reflects the threshold for statistical significance. The calculated p value for change in mealtime frequency is p = .84; Mean Difference (Final Values) = -.02

ADVERSE EVENTS:
Time Frame: Monitoring adverse events in children occurred across all study years through study completion, an average of 12 weeks from pre-test period, intervention period, post-test period for Phase 1 and an average of 24 weeks from pre-test period, intervention period, to post test period in Phase 2.
Description: The definitions did not differ from those described in clinicaltrials.gov
Arm/Group | Experimental: Phase 1 Usual Exposure | Experimental: Phase 1 Mealtime Support Activities | Experimental: Phase 2- Usual Exposure | Experimental: Phase 2- Meal Delivery and Receipt of Cookware
All-Cause Mortality (participants affected / at risk) | 0/434 | 0/65 | 0/152 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/434 | 0/65 | 0/152 | 0/159
Other Adverse Events (participants affected / at risk) | 0/434 | 0/65 | 0/152 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT02487251/Prot_SAP_000.pdf